CLINICAL TRIAL: NCT05733923
Title: Effectiveness of Papain-based Materials Compared With NaOCl-based Materials in Chemo-mechanical Caries Removal: A Randomized Controlled Trial
Brief Title: Evaluation of Chemo-mechanical Caries Removal Materials in Caries Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-OperativeDent-01-2023
Record Dates: First submitted 2023-01-29; First posted 2023-02-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries
Keywords: Chemo-mechanical caries removal; Papain-based agents; Minimum invasive dentistry; Conservative dentistry; Dental fear; Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Traditional excavation (Active Comparator): Mechanical caries Removal with low-speed Carbide Burs on a micromotor handpiece with air and water cooling.
  Interventions: Procedure: Traditional Escavation
- Sodium Hypochlorite CMCR (Experimental): chemomechanical caries removal using Sodium Hypochlorite Gel 2.5%.
  Interventions: Procedure: Excavation with Sodium Hypochlorite Gel 2.5%.
- Papacarie duo CMCR (Experimental): chemomechanical caries removal using Papacarie duo.
  Interventions: Procedure: Excavation with Papacarie Duo
- Selecti-solve CMCR (Experimental): chemomechanical caries removal using Selecti-solve Gel.
  Interventions: Procedure: Excavation with Brix3000
- Brix3000 CMCR (Experimental): chemomechanical caries removal using Brix3000.
  Interventions: Procedure: Excavation with Selecti-solve

INTERVENTIONS:
Procedure: Traditional Escavation — Patients will receive an operative procedure to remove dental caries by traditional excavation using Carbide burs on a micromotor handpiece at low speed with air and water cooling.
  - Group 6: 15 carious teeth will be excavated chemo-mechanically using Selecti-solve.
  Arms: Traditional excavation
Procedure: Excavation with Sodium Hypochlorite Gel 2.5%. — Patients will receive an operative procedure to remove dental caries by traditional excavation using Carbide burs on a micromotor handpiece at low speed with air and water cooling. In addition, teeth will be excavated chemo-mechanically using Sodium Hypochlorite Gel 2.5%.
  Arms: Sodium Hypochlorite CMCR
Procedure: Excavation with Papacarie Duo — Patients will receive an operative procedure to remove dental caries by traditional excavation using Carbide burs on a micromotor handpiece at low speed with air and water cooling. In addition, teeth will be excavated chemo-mechanically using a Papacarie Duo.
  Arms: Papacarie duo CMCR
Procedure: Excavation with Brix3000 — Patients will receive an operative procedure to remove dental caries by traditional excavation using Carbide burs on a micromotor handpiece at low speed with air and water cooling. In addition, teeth will be excavated chemo-mechanically using a Brix3000.
  Arms: Selecti-solve CMCR
Procedure: Excavation with Selecti-solve — Patients will receive an operative procedure to remove dental caries by traditional excavation using Carbide burs on a micromotor handpiece at low speed with air and water cooling. In addition, teeth will be excavated chemo-mechanically using a Selecti-solve.
  Arms: Brix3000 CMCR

SUMMARY:
• The evolution of conservative dentistry that adopts the preservation of tooth structure and affected dentin that can remineralize and save the pulp from exposure, in addition to pain and fear that companies' traditional caries removal methods had led to the development of chemomechanical caries removal materials (CMCR).

The old generations of CMCR agents were NaOcl-based materials which have disadvantages such as odor taste, Unpleasant smell, high cost, Limited shelf life, and time consumption.

• All of the reasons described led to a new generation of CMCR materials depending on Enzymes such as Papain.

Brix3000 and Papacarie duo are Papain-based materials with promising effects in caries removal and fewer disadvantages.

Selecti-solve is a dental gel whose active ingredient is papain enzyme, it removes dental caries without the need for anesthesia and is selective for the infected dentin layer only which avoids the unnecessary loss of dentin, enamel breaking, and pulp exposure.

This study aims to evaluate the efficacy of Papain-based materials compared to old NAOcl-Based materials in reducing the disadvantages of CMCR agents.

DETAILED DESCRIPTION:
In previous literature, there has not been any study that compared the whole group of chemo-mechanical caries removal materials with such a unique collection of Papain-based CMCR agents.

Papain-based agents could be promising materials in the evolution of Atraumatic Restorative treatment (ART) and Chemomechanical Caries removal methods that support conservative dentistry and the conservation of tooth structure and pulp vitality.

Brix3000 has EBE technology (Encapsulating Buffer Emulsion) that claims to elevate the efficiency of Papain Enzyme and permits the use of a higher concentration of Papain 3,000 U/mg in the whole material (10%).

Papacarie Duo has a unique combination of the main component of Papain Enzyme 6,000 U/mg and a small percentage of chloramine t that claims to increase efficiency and reduce the side effect of chloramine-based CMCR materials.

Selecti-solve is a new material that consists of Papain as the main product and has promising effects in chemo-mechanical caries removal methods.

ELIGIBILITY:
Inclusion Criteria:

* Wide carious lesion (Class 1 Black) on Molars at the middle third of dentine confirmed with a periapical x-ray
* No pulp involvement is assured with a periapical radiograph.
* Good oral hygiene
* Cooperated patient.
* No oral diseases.

Exclusion Criteria:

* Pulp exposure or bleeding during excavation.
* Pregnancy
* Systematic diseases
* Gingival and periodontal involvement.
* Lack of patient cooperation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Success in caries removal by a detecting dye | After procedure completion, which is expected to be within 20 minutes on average.
  The efficacy of caries removal will be assessed by a sharp probe aided by Caries Detector dye.
  The Cavity will be inspected after every application by a sharp probe to feel any tacky sensation in dentin, when it is all hard dentin, caries detector dye will be applied to aid the investigation.
  Caries detector dye will be left for 10 seconds and then rinsed with water, it will stain the organic matrix of less mineralized dentin so the cavity should be stained homogeneously so high-intensity colored spots refer to infected dentin and it will be removed.

SECONDARY OUTCOMES:
Time required for caries removal | After procedure completion, which is expected to be within 20 minutes on average.
  Time from the beginning of the caries excavation to the end of the process will be recorded in minutes using a stopwatch.
Pain perception during caries removal | After procedure completion, which is expected to be within 20 minutes on average.
  Visual analog scale (VAS) will be used to evaluate the pain perception during the procedure of caries removal.
  The patient will be asked to choose a number from 0 to 10 matching the intensity of his or her pain experience during the procedure.
  The higher the score, the more painful the procedure is.

CONTACTS AND LOCATIONS:
Overall Officials: Souad Abboud, DDS MSc PhD, Study Chair — Associate Professor of Restorative Dentistry, University of Damascus Faculty of Dentistry, Damascus; MHD Baraa Alsayed, DDS, Principal Investigator — MSc student, Department of Restorative Dentistry, University of Damascus, Damascus, Syria
Locations (1):
- Faculty of Dentistry, Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adham MM, El Kashlan MK, Abdelaziz WE, Rashad AS. Comparison of two minimally invasive restorative techniques in improving the oral health-related quality of life of pregnant women: a six months randomized controlled trial. BMC Oral Health. 2021 Apr 30;21(1):221. doi: 10.1186/s12903-021-01581-5. PMID 33931037
- [Background] AlHumaid J, Al-Harbi F, El Tantawi M, Elembaby A. X-ray microtomography assessment of Carisolv and Papacarie effect on dentin mineral density and amount of removed tissue. Acta Odontol Scand. 2018 May;76(4):236-240. doi: 10.1080/00016357.2017.1406614. Epub 2017 Nov 21. PMID 29161950
- [Background] Cardoso M, Coelho A, Lima R, Amaro I, Paula A, Marto CM, Sousa J, Spagnuolo G, Marques Ferreira M, Carrilho E. Efficacy and Patient's Acceptance of Alternative Methods for Caries Removal-a Systematic Review. J Clin Med. 2020 Oct 23;9(11):3407. doi: 10.3390/jcm9113407. PMID 33114249
- [Background] de Souza TF, Martins ML, Tavares-Silva CM, Fonseca-Goncalves A, Maia LC. Treatment time, pain experience and acceptability of the technique for caries removal in primary teeth using the ART approach with or without Brix3000 papain gel: a preliminary randomised controlled clinical trial. Eur Arch Paediatr Dent. 2022 Oct;23(5):777-785. doi: 10.1007/s40368-021-00669-4. Epub 2021 Oct 2. PMID 34599744
- [Background] Divya G, Prasad MG, Vasa AA, Vasanthi D, Ramanarayana B, Mynampati P. Evaluation of the Efficacy of Caries Removal Using Polymer Bur, Stainless Steel Bur, Carisolv, Papacarie - An Invitro Comparative Study. J Clin Diagn Res. 2015 Jul;9(7):ZC42-6. doi: 10.7860/JCDR/2015/12705.6202. Epub 2015 Jul 1. PMID 26393204
- [Background] Santos TML, Bresciani E, Matos FS, Camargo SEA, Hidalgo APT, Rivera LML, Bernardino IM, Paranhos LR. Comparison between conventional and chemomechanical approaches for the removal of carious dentin: an in vitro study. Sci Rep. 2020 May 15;10(1):8127. doi: 10.1038/s41598-020-65159-x. PMID 32415190
- [Background] Katiyar A, Gupta S, Gupta K, Sharma K, Tripathi B, Sharma N. Comparative Evaluation of Chemo-mechanical and Rotary-mechanical Methods in Removal of Caries with Respect to Time Consumption and Pain Perception in Pediatrc Dental Patients. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):115-119. doi: 10.5005/jp-journals-10005-1896. PMID 34326596
- [Background] Mancini L, Pisaneschi A, Mancini V, Ginoble M, Quinzi V, Marchetti E, Marzo G. BRIX3000(R) Papain Gel for Cavity Treatment in the Adult Patient. Case Rep Dent. 2021 Jun 12;2021:6624825. doi: 10.1155/2021/6624825. eCollection 2021. PMID 34194848
- [Background] Matsumoto SF, Motta LJ, Alfaya TA, Guedes CC, Fernandes KP, Bussadori SK. Assessment of chemomechanical removal of carious lesions using Papacarie Duo: randomized longitudinal clinical trial. Indian J Dent Res. 2013 Jul-Aug;24(4):488-92. doi: 10.4103/0970-9290.118393. PMID 24047844